CLINICAL TRIAL: NCT00413400
Title: Effects of Etanercept in Patients With the Metabolic Syndrome (II)
Brief Title: Study of TNF-Antagonism in the Metabolic Syndrome (II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Steven Grinspoon, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-P-001060
Record Dates: First submitted 2006-12-07; First posted 2006-12-19 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Metabolic Syndrome
Keywords: Inflammation; Visceral adiposity; TNF; Adiponectin; glucose tolerance; endothelial function; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Etanercept (Active Comparator)
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — 50 mg one syringe sc 2X per week for three months followed by 50 mg one syringe sc 1X per week for three months
  Other Names: Enbrel
  Arms: Etanercept
Drug: Placebo — 50 mg one syringe sc 2x per week for three months followed by 50 mg one syringe sc 1X per week for three months
  Arms: Placebo

SUMMARY:
This study will investigate whether etanercept will result in improved inflammatory indices, glucose tolerance and endothelial function in patients with the metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome is an increasingly prevalent disorder associated with elevated risks of type II DM (diabetes mellitus) and cardiovascular morbidity and mortality. A subclinical inflammatory state is thought to contribute to the pathophysiology of metabolic syndrome, insulin resistance, and coronary artery disease (CAD). Tumor Necrosis Factor (TNF) -alpha is an inflammatory cytokine that is increased in a spectrum of inflammatory diseases as well as in insulin resistance. TNF-alpha antagonists are clinically effective in the inflammation of arthritides, and have recently been shown by our group to decrease inflammatory cardiovascular risk markers in metabolic syndrome. Data suggests that adiponectin, a recently discovered adipocytokine that may protect against the development of insulin resistance and atherosclerosis, may be downregulated by TNF-alpha. In addition, population based studies have shown that those with the highest levels of TNF-alpha have an increased relative risk of cardiovascular morbidity while rheumatoid arthritis patients treated with TNF-alpha blockade appear protected from cardiovascular disease. We will perform a 6-month study in which we will administer etanercept, a TNF-alpha receptor fusion protein, to subjects with metabolic syndrome to investigate its effect on surrogate markers of cardiovascular disease, including inflammatory markers, adiponectin and glucose tolerance and endothelial function. The results of the proposed study will have broad implications regarding the physiological role of TNF-alpha on the inflammatory cascade, cardiovascular indices and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

1. Hyperinsulinemia in the upper quartile of the non-diabetic population defined as >= 10 mU/mL (based on Framingham Data, oral communication, James Meigs, MD) or fasting glucose 110-126 mg/dL
2. Plus two of the following:

   * Abdominal obesity defined by waist hip ratio > 0.90 for men and > 0.85 for women and BMI > 30 kg/m2
   * Dyslipidemia including serum triglycerides >= 150 mg/dl or serum high density lipoprotein (HDL) < 0.9 mmol/L for men (35 mg/dL) and < 1.0 mmol/L (39mg/dL) for women
   * Hypertension defined as blood pressure >= 140/90 or on medication

Exclusion Criteria:

1. Age < 18 or > 60 years
2. Body mass index (BMI) < 30 kg/m2
3. Positive tuberculosis (purified protein derivative [PPD]) skin test (5mm induration or more) on screening
4. Mycobacterial disease treated less than 6 months.
5. Current or recurrent infection or any underlying condition that may predispose to infection or anyone who has been admitted to the hospital due to bacteremia, pneumonia or any other serious infection.
6. Therapy with glucocorticoid or immunosuppressant at time of recruitment or within past 3 months.
7. Prior or concurrent cyclophosphamide therapy
8. Use of a live vaccine 90 days prior to, or during this study.
9. History of blood dyscrasia including any kind of anemia, thrombocytopenia, pancytopenia. Women with a reversible cause of anemia that has resolved will be eligible.
10. Hemoglobin < 11 g/dl
11. History of malignancy (except patients with surgically cured basal cell or squamous cell skin cancers who will be eligible)
12. History of organ transplantation
13. HIV-positive status determined by HIV test at screening or known history of any other immuno-suppressing disease.
14. Hepatitis B or hepatitis C infection detected at screening, lupus (SLE), history of multiple sclerosis, transverse myelitis, optic neuritis or epilepsy
15. Patients with known autoimmune or inflammatory conditions (excluding patients with stable, treated hypothyroidism)
16. Severe comorbidities (diabetes mellitus requiring insulin, congestive heart failure (CHF) (EF<50% at baseline will be exclusionary) of any severity, myocardial infarction (MI), cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 3 months of screening visit, unstable angina pectoris, oxygen-dependent severe pulmonary disease
17. Uncontrolled systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg
18. Fasting blood glucose > 126 mg/dL
19. Creatinine > 1.5
20. Current use of insulin, any oral anti-hyperglycemic agents (including insulin sensitizing agents). Initiation of insulin, oral hypoglycemics, or insulin sensitizing agents during the study will result in discontinuation from the study.
21. Initiation of statins, niacin, antihypertensive or fibrate therapy within 6 weeks of the study. Chronic use of fibrates, niacin, or antihypertensives for > 6 weeks prior to study initiation at a stable dose is not exclusionary, but chronic use of statins for > 6 months is exclusionary. Initiation of statins, fibrates, niacin or antihypertensive treatments during the study is not exclusionary but will be considered in the analysis (see Protection against risks).
22. Positive pregnancy test or lactating females
23. Women of child-bearing potential not currently using non-hormonal birth control methods including barrier methods (intrauterine device [IUD], condoms, diaphragms) or abstinence
24. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
25. Subjects who have known hypersensitivity to Enbrel or any of its components or who is known to have antibodies to etanercept
26. Concurrent sulfasalazine therapy
27. History of recent alcohol or substance abuse (< 1 year)
28. Any condition judged by the patient's physician to cause this clinical trial to be detrimental to the patient.
29. History of non-compliance with other therapies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, Principal Investigator — MGH
Locations (1):
- MGH, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 12/2006 to 3/2009
Groups:
- Placebo: Placebo injections, subcutaneously, twice weekly x 3 months, then once weekly x 3 months
- Etanercept: Etanercept 50mg subcutaneously twice weekly x 3 months, then once weekly x 3 months
Period: Overall Study
Arm/Group | Placebo | Etanercept
Started | 24 | 16
3 Month Visit | 22 | 12
Completed | 22 | 12
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etanercept | Total
Number analyzed (Participants) | 24 | 16 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 16 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (8) | 41 (9) | 45 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 12 | 8 | 20
Region of Enrollment [Number; unit: participants]
  United States | 24 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: C-reactive Protein (CRP)
Description: As a measure of C-reactive protein (CRP), which is an inflammatory marker, Log10 of the CRP at 6 months is reported
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Log10 mg/L
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
Log10 mg/L | 0.61 (0.06) | 0.68 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; treatment effect (etanercept vs. placebo) using ANCOVA including baseline CRP, age, and race; Test type: Superiority or Other; p = 0.20, ANCOVA

2. Primary Outcome: Interleukin-6 (IL-6)
Description: 6 month value of IL-6 (pg/mL)
Time Frame: 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
pg/mL | 8.2 (1.1) | 11.3 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; within subject percent changes calculated for each timepoint and repeated measures ANCOVA controlling for age and race performed; Test type: Superiority or Other; p = 0.92, Repeated Measures ANCOVA

3. Primary Outcome: Adiponectin
Description: The ratio of circulating high molecular weight (HMW) adiponectin to total adiponectin ratio (HMW:total Adiponectin) at 6 months is reported.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: (ratio)
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
(ratio) | 0.30 (0.08) | 0.40 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; within subject percent changes were calculated for each time point, then repeated measures ANCOVA controlling for age and race performed; Test type: Superiority or Other; p = 0.02, Repeated Measures ANCOVA

4. Secondary Outcome: Glucose Tolerance
Description: Fasting glucose (mg/dL) at 6mo
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
mg/dL | 95 (5) | 91 (6)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; percent change calculated then repeated measures ANCOVA performed controlling for age and race; Test type: Superiority or Other; p = 0.02, repeated measures ANCOVA

5. Secondary Outcome: Endothelial Function
Description: Reactive Hyperemia Index (RHI) using peripheral artery tonometry (using Endo-PAT 2000). Peripheral artery tonometry measures blood flow in the tip of the index finger at baseline and in response to vaso-occlusion (inflated blood pressure cuff). The reactive hyperemia index is an index of vasodilation after occlusion compared to baseline. A higher value indicates better vasoreactivity. As this is a relatively new test, there are no thoroughly validated clinically utilized norms.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: (index)
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
(index) | 1.8 (0.11) | 2.0 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; ANCOVA controlling for baseline value, age, race; Test type: Superiority or Other; p = 0.46, ANCOVA

6. Secondary Outcome: White Blood Cell (WBC) Count
Description: Change in WBC during study (WBC at six months minus WBC at baseline)
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: th/cumm
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
th/cumm | -0.17 (0.23) | -0.04 (0.45)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority or Other; p = 0.78, t-test, 2 sided

7. Secondary Outcome: Cardiac Echo Ejection Fraction (EF)
Description: change in EF (6mo - baseline). Please note that the value given is the absolute change in EF (which has units of percent), not the percent change in the variable.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: percent
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
percent | 1.1 (0.7) | -1.1 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority or Other; p = 0.11, t-test, 2 sided

8. Secondary Outcome: Body Composition
Description: 6 month visceral adipose tissue (cm^2) - cross-sectional area of the visceral adipose tissue at the level of the 4th lumbar vertebrae was measured using single-slice abdominal computed tomography (CT) scan
Time Frame: 6 months
Measure: Mean (Standard Error); unit: cm^2
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
cm^2 | 206 (18) | 186 (14)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; ANCOVA controlling for baseline value, age, race; Test type: Superiority or Other; p = 0.59, ANCOVA

9. Secondary Outcome: Tumor Necrosis Factor (TNF) Receptor
Description: Circulating concentrations of Tumor necrosis factor receptor 2 (TNFR2) at 6 months
Time Frame: 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
pg/mL | 2573 (148) | 4518 (329)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; within subject percent changes calculated then repeated measures ANCOVA controlling for age and race performed; Test type: Superiority or Other; p < 0.0001, Repeated measures ANCOVA

10. Secondary Outcome: Other Adipocytokines
Description: circulating resistin at 6 months
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
ng/mL | 6.7 (0.5) | 8.6 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; within subject percent changes calculated then repeated measures ANCOVA performed controlling for age and race; Test type: Superiority or Other; p = 0.08, Repeated Measures ANCOVA

11. Secondary Outcome: Lipid Levels
Description: total cholesterol (mg/dL) at 6 months
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 22 | 12
mg/dL | 196 (9) | 201 (12)
Statistical Analysis 1: Comparison: Placebo vs Etanercept; ANCOVA controlling for baseline value, age, and race; Test type: Superiority or Other; p = 0.55, ANCOVA

12. Secondary Outcome: Adipocyte Messenger Ribonucleic Acid (mRNA) Levels of Adipocytokines Including Tumor Necrosis Factor (TNF) -Alpha
Description: fold-change in subcutaneous adipose tissue expression of TNF-alpha (mRNA) after 6 months
Time Frame: 6 months
Measure: Mean (Standard Error); unit: fold-change
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 8 | 4
fold-change | 2.3 (0.7) | 1.1 (0.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Etanercept
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/16
Other Adverse Events (participants affected / at risk) | 8/24 | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Etanercept (N=16)
Operative Surgical Procedure (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — 1 placebo subject had surgery for cervical disc repair, and 1 etanercept subject had planned (elective) knee surgery
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) — 1 subject receiving etanercept developed transient parasthesia in leg after giving study medication. Study drug was discontinued and symptoms resolved.
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) — Exacerbation of pre-existing schizophrenia requiring hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Etanercept (N=16)
Bakers Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dental Infection (Infections and infestations) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Foot Swelling (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leukocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) — Mild intermittent symptoms of tingling in hands and feet in a subject who had also experienced these symptoms prior to study participation
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No